CLINICAL TRIAL: NCT06907797
Title: Tools for Reducing Inequity in Acute Leukemia (TRIAL): Beta Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: American Society of Clinical Oncology (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrew Hantel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-698; K08CA273043 (NIH)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acute Leukemia; Leukemia
Keywords: Acute Leukemia; Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TRIAL Web-Based Application (Experimental): Enrolled participants will complete:
  * Baseline visit and questionnaires
  * Access to web application over the course of 14 days.
  * End of study questionnaires
  * 12 participants will take part in semi-structured interviews with study staff which will be audio recorded.
  Interventions: Behavioral: TRIAL Web-Based Application

INTERVENTIONS:
Behavioral: TRIAL Web-Based Application — A web-based application that provides disease and trial education and access to resources provided by the Leukemia and Lymphoma Society (LLS). iPads will be provided to participants for 14 days.
  Other Names: TRIAL

SUMMARY:
This study aims to test the Tools for Reducing Inequity in Acute Leukemia (TRIAL) web-based application that is designed to support participants with acute leukemia by providing information and resources about leukemia and clinical trial participation.

DETAILED DESCRIPTION:
The goal of this single-arm pilot study is to test the TRIAL web application which is designed to reduce inequity in clinical trial enrollment among participants with acute leukemia. The application aims to facilitate access to clinical trials and reduce barriers for underrepresented groups.

The research study procedures include screening for eligibility and questionnaires.

Participation in this research study is expected to last about 14 weeks.

It is expected about 75 people will participate in this study.

The National Cancer Institute (NCI) and American Society of Clinical Oncology (ASCO) are providing funding for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* English speaking
* Ability to understand and willingness to sign written informed consent
* Clinical suspicion of acute leukemia
* Admitted to DFCI-affiliated inpatient unit

Exclusion Criteria:

* Cognitive impairment rendering the individual unable to participate in beta testing

  * This will be assessed by focused chart review and consultation with the patients' inpatient care team.
* The following populations will be excluded: adults unable to consent, individuals who are not yet adults (infants, children, teenagers <18 years old), prisoners.
* Inability to participate in in-person application testing.
* Patients who participated in alpha-testing through protocol 23-404 (Appendix A)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Post-Test Completion Rate | Day 14 or date of discharge
  Defined as the proportion of completed post-tests compared to the overall total of 75. Retention feasibility is defined as ≥ 70% of post-test completions, or 53 completions.
System Usability Scale (SUS) Score | Day 14 or date of discharge
  Assessed by the System Usability Scale (SUS), a 10-item measure rated on a 5-point Likert scale from 1 "Strongly Disagree" to 5 "Strongly Agree" with a total scores range of 0 to 100. A higher score represents greater usability.
Percentage of Participants Scoring ≥68 on SUS | approximately 12 months (based on total accrual duration)
  Defined as the proportion of participants who score ≥68 on the SUS compared to the overall enrollment of 75 participants. Usability of the intervention is defined as >70%, or 53 participants.

SECONDARY OUTCOMES:
Participant Screening Rate | approximately 12 months (based on total accrual duration)
  Defined as the proportion of enrollees over the number of participants approached for study enrollment.
Participant Eligibility Rate | approximately 12 months (based on total accrual duration)
  Defined as the proportion of enrollees over the number of participants eligible for study enrollment.
Change in Seven-Item Knowledge Scale (SIKS) Score from Baseline to Post-Test | Baseline and day 14 or date of discharge (post-test)
  Assessed by the Seven-Item Knowledge Scale (SIKS) which is comprised of items covering general clinical research statements. Respondents indicate whether a statement is "True," "False," or "Don't know." Scoring is based on the number of correct items (range 0-100). "Don't know" and omitted responses do not count toward the score. A score of 70 or higher indicates adequate knowledge.
Change in Attitudes to Randomized Trials Questionnaire (ARTQ) Score from Baseline to Post-Test | Baseline and day 14 or day of discharge (post-test)
  Assessed by the Attitudes to Randomized Trials Questionnaire (ARTQ), a 7-item measure with answers of "Yes, "No," or "Do Not Know." The first three items represent willingness to participate in a clinical trial. These items will be assigned a value of 1 for an answer of "Yes" or 0 for an answer of "No or Do Not Know" and summed to obtain overall willingness. Change = (Day 14 or Discharge score - Baseline score)/Baseline score
Change in Trust in Medical Researchers Scale (TMRS) Score from Baseline to Post-Test | Baseline and day 14 or day of discharge (post-test)
  Assessed by the Trust in Medical Researchers scale (TMRS), a 12-item measure rated on a 5-point Likert scale with answers ranging from 1 "Strongly Disagree" to 5" Strongly Agree" with a total scores range of 12 to 48. A higher score indicates greater trust in medical researchers.
Ottawa Preparation for Decision Making Scale (Prep-DM) Score | Day 14 or date of discharge
  Assessed by the Ottawa Preparation for Decision Making Scale (Prep-DM), a 10-item measure rated on a 5-point Likert scale with answers ranging from 1 "Not at All" to 5 "A Great deal" with a total scores range of 0 to 100. A higher score indicates higher perceived level of preparedness for decision making.
Acceptability of Intervention Measure (AIM) Score | Day 14 or date of discharge
  Assessed by the Acceptability of Intervention Measure (AIM), a 4-item measure rated on a 5-point Likert scale with answers ranging from 1 "Completely disagree" to 5 "Completely agree." A total scores range is 4 to 20 with a higher score indicating greater acceptability.
Participant Enrollment Agreement Rate | approximately 12 months (based on total accrual duration)
  Defined as the proportion of participants that agree to participate in a clinical trial divided by the number of enrollment opportunities. For the purposes of this study, which does not impact clinician behaviors or trial eligibility criteria, a patient who agrees to enroll in a study is someone who is presented with information about a study and agrees to participate and either screen fails or passes screening and consents to participate. An enrollment opportunity is defined as a patient who is identified by the care team as screen eligible for a clinical trial and approached for participation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hantel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu